CLINICAL TRIAL: NCT00105274
Title: Intermediate Phenotype and Genetic Mechanisms for Psychosis and Cognitive Disturbance in 22q11.2-Hemideletion Syndrome
Brief Title: Velocardiofacial (VCFS; 22q11.2; DiGeorge) Syndrome Study
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050110; 05-M-0110
Record Dates: First submitted 2005-03-10; First posted 2005-03-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-02

CONDITIONS: DiGeorge Syndrome; Velocardiofacial Syndrome; 22q11.2 Syndrome
Keywords: Velocardiofacial Syndrome; Susceptibility Genes; Neuroimaging; 22q11.2; Psychosis; Mircodeletion; DiGeorge Syndrome; 22q11.2 Syndrome
MeSH Terms: conditions — DiGeorge Syndrome; Psychotic Disorders

SUMMARY:
Velocardiofacial syndrome, also known as 22q11.2 syndrome or DiGeorge syndrome, has been associated with many features such as a cleft palate, heart defects, and learning, speech and feeding problems. It is caused by the absence of a number of genes on chromosome 22, but the mechanism by which this inborn abnormality causes the clinical problems is not known.

In this study by the National Institute of Mental Health and the Office of Rare Diseases, we are recruiting participants with 22q11.2 syndrome to come for a three-day stay to our main campus in Bethesda, MD, to participate in a study in which we will investigate the genetic makeup of their cells together with several studies of brain function with advanced research imaging. The goal of this study is to understand how the genes missing in 22q11.2 syndrome are related to the increased occurrence of psychiatric problems, such as psychosis, in this syndrome. Participants must be 18-50 years of age, have some high school education and not currently be taking antipsychotic medication. Travel costs to Bethesda for participants and an accompanying person will be paid, and participants are reimbursed for their time in participating in the study. A blood draw is required. All research procedures have been designated as "minimal risk" procedures.

...

DETAILED DESCRIPTION:
22q11.2 (DiGeorge MIM#188400, Velocardiofacial MIM#192430) syndrome is a hemizygous microdeletion on 22q11.2 of typically 3Mb, encompassing approximately 30 genes and mediated by aberrant homologous recombination and unequal crossing-over events between intrachromosomal flanking low-copy repeats (LCRs). The incidence is 1:4000 live births. While somatic symptoms include congenital cardiovascular and craniofacial abnormalities, recurrent infections and hypocalcemia1 , the most prevalent group of symptoms are neuropsychiatric and include cognitive dysfunction with mild mental retardation, behavioral difficulties and psychosis. The syndrome is associated with a lifetime prevalence of schizophrenia-like illness (phenotypically mostly similar to sporadic schizophrenia) of approximately 25 times that of the general population making the presence of this hemideletion the strongest known risk factor for the development of schizophrenia excepting the presence of a monozygotic twin with the illness. The 22q11 region is implicated in the risk architecture of schizophrenia by several linkage studies and harbors a number of proposed susceptibility genes including genes for Catechol-O-methyltransferase (COMT), proline dehydrogenase (PRODH) and ZDHHC8. The neural basis of these pronounced neurocognitive and psychiatric abnormalities is unknown. The present work proposes to (a) study a group of exceptionally high-functioning, normal intelligence, psychosis-free individuals with 21q11.2 syndrome using a hierarchical multimodal imaging approach to define the intermediate systems level phenotype of the disease combined with deletion mapping techniques and (b) to study the functional effects of single nucleotide polymorphisms in genes in the hemideleted region that have been implicated in schizophrenia, taking advantage of the unique fact that the hemizygous deletion allows immediate construction of molecular haplotypes and of potential epistatic allelic effects. This work is expected to (a) elucidate the pathophysiology of the CNS manifestations of the 22q11.2 syndrome and yield a brain intermediate phenotype that will allow studies in small and atypical deletion individuals in an effort to define individual genes responsible for neurocognitive deficit and increased risk for psychosis, (b) facilitate the identification of functional mechanisms underlying increased risk for schizophrenia for individual susceptibility genes in the deletion and for interacting risk alleles within the deleted locus and (c) prepare the ground for a clinical protocol in which the results from (a) and (b) can be applied to a prospective study evaluating early diagnostic and interventional approaches based on genetic risk and intermediate phenotype ascertainment in this group of patients at high risk for the development of psychosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Only adults between age 18 and 50 will be studied. 22q11.2 participants: 22q11.2 deletion will be confirmed by FISH. IQ (WAIS). In phase 1: IQ in the general range of the population (greater than 85) as ascertained using the 2- and 4-subset forms of the Wechsler Abbreviated Scale of Intelligence (Wechsler, 1999). Informed consent.

EXCLUSION CRITERIA:

(Phase 1 only) Any lifetime diagnosis of schizophrenia, schizoaffective disorder, or schizotypal disorder and/or current pychotropic medication or any neuroleptic medication in the previous year. (all phases) Chronological age greater 50 years. Contraindication of MRI scanning (ferromagnetic metal implanted in body, prostheses containing such metal, pacemaker devices). Pregnancy. Medication affecting central nervous function. Severe somatic disorders precluding travel to the clinical center or participation in imaging procedures. Hypothyroidism not compensated by medication. Neurological disorders excluding those of exclusively peripheral location.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2005-03-07; Study Completion 2010-02-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lindsay EA. Chromosomal microdeletions: dissecting del22q11 syndrome. Nat Rev Genet. 2001 Nov;2(11):858-68. doi: 10.1038/35098574. PMID 11715041
- [Background] Edelmann L, Pandita RK, Spiteri E, Funke B, Goldberg R, Palanisamy N, Chaganti RS, Magenis E, Shprintzen RJ, Morrow BE. A common molecular basis for rearrangement disorders on chromosome 22q11. Hum Mol Genet. 1999 Jul;8(7):1157-67. doi: 10.1093/hmg/8.7.1157. PMID 10369860
- [Background] Botto LD, May K, Fernhoff PM, Correa A, Coleman K, Rasmussen SA, Merritt RK, O'Leary LA, Wong LY, Elixson EM, Mahle WT, Campbell RM. A population-based study of the 22q11.2 deletion: phenotype, incidence, and contribution to major birth defects in the population. Pediatrics. 2003 Jul;112(1 Pt 1):101-7. doi: 10.1542/peds.112.1.101. PMID 12837874